CLINICAL TRIAL: NCT01925287
Title: Novel Strategies for the Enhancement of the Potency of Nutraceuticals With Low Oral Bioavailability and Their Application in Novel Functional Foods for Optimum Protection of the Aging Brain
Brief Title: Oral Bioavailability of Curcumin From Micronized Powder and Liquid Micelles in Healthy Young Women and Men
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 01EA1334AHS1
Record Dates: First submitted 2013-08-13; First posted 2013-08-19 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Pharmacokinetics of Novel Curcumin Formulations; Safety of Novel Curcumin Formulations
Keywords: bioavailability; curcumin; curcuma longa; healthy humans; safety; sex differences
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Native curcumin powder (Active Comparator): 500 mg curcumin as native powder
  Interventions: Dietary Supplement: curcumin
- Micronized curcumin powder (Experimental): 500 mg curcumin as micronized powder
  Interventions: Dietary Supplement: curcumin
- Curcumin micelles (Experimental): 500 mg curcumin incorporated into liquid micelles
  Interventions: Dietary Supplement: curcumin

INTERVENTIONS:
Dietary Supplement: curcumin — 500 mg curcumin were given orally either as native powder, micronized powder, or liquid micelles

SUMMARY:
Background: The oral bioavailability of curcumin is low due to its limited intestinal uptake, rapid metabolism and excretion from the body. Considering its potent reported health-beneficial properties, researchers have tried to increase its bioavailability as a means to enhance its biological activities.

Objective: The aim of the project was to develop novel curcumin formulations with enhanced oral bioavailability and to study the safety of the formulations and potential sex-differences in humans.

Design: In this single-blind crossover study with three arms separated by ≥1-week washout periods, healthy subjects (13 women, 10 men) were provided standardized meals and took, in random order, a single oral dose of 500 mg curcumin as native powder, micronized powder, or liquid micelles. Blood and urine samples were collected in intervals for 24 h and total curcumin, demethoxycurcumin, and bis-demethoxycurcumin were quantified.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with routine blood chemistry values within the normal ranges

Exclusion Criteria:

* overweight (BMI >30 kg/m2)
* metabolic and endocrine diseases
* pregnancy
* lactation
* drug abuse
* use of dietary supplements or any form of medication (with the exception of oral contraceptives)
* smoking
* frequent alcohol consumption (>20 g ethanol/d)
* adherence to a restrictive dietary regimen
* physical activity of more than 5 h/wk
* participation in a clinical trial within the past 3 months prior to recruitment
* known intolerance against curcuma

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of total curcumin [nmol/L*h] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total curcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Area under the plasma concentration versus time curve (AUC) of total demethoxycurcumin [nmol/L*h] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total demethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Area under the plasma concentration versus time curve (AUC) of total bisdemethoxycurcumin [nmol/L*h] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total bisdemethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Maximum plasma concentration (Cmax) of total curcumin [nmol/L] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total curcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Maximum plasma concentration (Cmax) of total demethoxycurcumin [nmol/L] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total demethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Maximum plasma concentration (Cmax) of total bisdemethoxycurcumin [nmol/L] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total bisdemethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total curcumin [h] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total curcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total demethoxycurcumin [h] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total demethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total bisdemethoxycurcumin [h] | 0, 0.5, 1, 1.5, 2, 4, 6, 8 and 24 h post-dose
  Total bisdemethoxycurcumin was determined after deconjugation with beta-glucuronidase/sulphatase

SECONDARY OUTCOMES:
Serum aspartate transaminase activity [U/L] | Baseline
Serum aspartate transaminase activity [U/L] | 4 h post-dose
Serum aspartate transaminase activity [U/L] | 24 h post-dose
Serum alanine transaminase activity [U/L] | Baseline
Serum alanine transaminase activity [U/L] | 4 h post-dose
Serum alanine transaminase activity [U/L] | 24 h post-dose
Serum gamma-glutamyl transferase activity [U/L] | Baseline
Serum gamma-glutamyl transferase activity [U/L] | 4 h post-dose
Serum gamma-glutamyl transferase activity [U/L] | 24 h post-dose
Serum alkaline phosphatase activity [U/L] | Baseline
Serum alkaline phosphatase activity [U/L] | 4 h post-dose
Serum alkaline phosphatase activity [U/L] | 24 h post-dose
Serum bilirubin [mg/dL] | Baseline
Serum bilirubin [mg/dL] | 4 h post-dose
Serum bilirubin [mg/dL] | 24 h post-dose
Serum uric acid [mg/dL] | Baseline
Serum uric acid [mg/dL] | 4 h post-dose
Serum uric acid [mg/dL] | 24 h post-dose
Serum cystatin C [mg/L] | Baseline
Serum cystatin C [mg/L] | 4 h post-dose
Serum cystatin C [mg/L] | 24 h post-dose
Glomerular filtration rate [mL/min] | Baseline
Glomerular filtration rate [mL/min] | 4 h post-dose
Glomerular filtration rate [mL/min] | 24 h post-dose
Serum creatinine [mg/dL] | Baseline
Serum creatinine [mg/dL] | 4 h post-dose
Serum creatinine [mg/dL] | 24 h post-dose
Serum total cholesterol [mg/dL] | Baseline
Serum total cholesterol [mg/dL] | 4 h post-dose
Serum total cholesterol [mg/dL] | 24 h post-dose
Serum HDL cholesterol [mg/dL] | Baseline
Serum HDL cholesterol [mg/dL] | 4 h post-dose
Serum HDL cholesterol [mg/dL] | 24 h post-dose
Serum LDL cholesterol [mg/dL] | Baseline
Serum LDL cholesterol [mg/dL] | 4 h post-dose
Serum LDL cholesterol [mg/dL] | 24 h post-dose
Serum triacylglycerols [mg/dL] | Baseline
Serum triacylglycerols [mg/dL] | 4 h post-dose
Serum triacylglycerols [mg/dL] | 24 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Ph.D., Principal Investigator — University of Hohenheim, Stuttgart, Germany
Locations (1):
- University of Hohenheim, Stuttgart, Germany

REFERENCES:
- [Result] Schiborr C, Kocher A, Behnam D, Jandasek J, Toelstede S, Frank J. The oral bioavailability of curcumin from micronized powder and liquid micelles is significantly increased in healthy humans and differs between sexes. Mol Nutr Food Res. 2014 Mar;58(3):516-27. doi: 10.1002/mnfr.201300724. Epub 2014 Jan 9. PMID 24402825
- See also: Website of the research group — http://www.nutrition-research.de/